CLINICAL TRIAL: NCT03691363
Title: Mobile Subthreshold Exercise Program (M-STEP) for Concussion
Brief Title: Mobile Subthreshold Exercise Program for Concussion
Acronym: M-STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Sara PD Chrisman, MD MPH, Assistant Professor, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00001039
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Brain Concussion
Keywords: child; Adolescent; exercise; rehabilitation; physical activity; virtual; mobile health
MeSH Terms: conditions — Brain Concussion; Motor Activity | interventions — SE 1-step Futurabond M

STUDY DESIGN:
Intervention Model Description: All youth will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M-STEP (Experimental): Mobile exercise intervention
  Interventions: Behavioral: M-STEP

INTERVENTIONS:
Behavioral: M-STEP — Youth will be assessed using actigraphy at baseline, and will then be asked to exercise for 1) a duration of 10 minutes > MVPA at baseline with 2) HR>120 while being monitored by a Fitbit. Youth will be asked to exercise daily, and intensity and duration will be increased every few days for a goal of 60 minutes per day at a HR>140 (low end of MVPA). The intervention will be 6 weeks in duration.
  Other Names: Sub-threshold exercise

SUMMARY:
Non-randomized pilot intervention using mobile-administered sub-threshold exercise to treat youth with prolonged symptoms of concussion.

DETAILED DESCRIPTION:
6-week pilot study of a novel intervention for concussion, administering a sub-threshold exercise program in a mobile fashion using video conferencing and providing feedback using wrist-worn accelerometry and heart rate monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Concussion diagnosed by a healthcare provider that occurred 2 weeks-6 months ago
* Continued symptoms with at least 3 symptoms on the HBI and a score of 20+
* No other issues that would preclude physical activity
* Parents and youth are English-speaking

Exclusion Criteria:

- Already participating in >30 minutes of MVPA/day

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Health Behavior Inventory (HBI), 21 item 0-3 likert, higher scores indicate more severe symptoms | Trajectory over 6 weeks (baseline, 3 weeks, 6 weeks)
  Self-report questionnaire regarding concussive symptoms

SECONDARY OUTCOMES:
Change in Pediatric Quality of Life Inventory (PedsQL), 23 item 0-4 likert, converted to a 0-100 scale, higher scores indicate improved function | Trajectory over 6 weeks (baseline, 3 weeks, 6 weeks)
  Self-report questionnaire regarding Health-related quality of life
Change in Fear of pain questionnaire (FOPQ)-P/C, adapted for concussion, 24 item (child) and 23 item (parent) 0-4 likert, higher scores indicate greater fear-avoidance | Trajectory over 6 weeks (baseline, 3 weeks, 6 weeks)
  Self-report questionnaire completed by parent and child regarding their fear of concussive symptoms and avoidance of activities that might produce concussive symptoms
Change in Patient Health Questionnaire 9 (PHQ-9), 9 item 0-3 likert, higher scores indicate greater symptoms | Trajectory over 6 weeks (baseline, 3 weeks, 6 weeks)
  Self-report questionnaire of depression symptoms
Change in Adolescent Sleep Wake Scale (ASWS), 10-item 0-5 likert, higher scores indicate improved sleep quality | Trajectory over 6 weeks (baseline, 3 weeks, 6 weeks)
  Self-report 10-item questionnaire regarding difficulty falling asleep, night wakenings and other sleep issues
Change in Generalized anxiety disorder--7 item (GAD7), 7-item 0-3 likert, higher scores indicate more severe symptoms | Trajectory over 6 weeks (baseline, 3 weeks, 6 weeks)
  Self-report questionnaire regarding anxiety symptoms (7-item)
Study Satisfaction Questionnaire | 6 weeks
  8 item survey regarding satisfaction with study, 0-3 likert, higher scores indicate greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Sara PD Chrisman, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Chrisman SPD, Mendoza JA, Zhou C, Palermo TM, Gogue-Garcia T, Janz KF, Rivara FP. Pilot Study of Telehealth Delivered Rehabilitative Exercise for Youth With Concussion: The Mobile Subthreshold Exercise Program (MSTEP). Front Pediatr. 2021 May 28;9:645814. doi: 10.3389/fped.2021.645814. eCollection 2021. PMID 34123963